CLINICAL TRIAL: NCT00613301
Title: Pramipexole Special Survey on Patients Without Concomitant Use of L-Dopa
Brief Title: Special Survey on Parkinson's Disease (PD) Patients Without Concomitant Use of L-Dopa
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.549
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-11-23 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The survey is conducted to collect safety and effectiveness information in Parkinson's Disease patients treated with Pramipexole without concomitant L-Dopa supplementation in the daily clinical settings in Japan.

ELIGIBILITY:
Inclusion Criteria:

Patients with Parkinson's disease who do not receive L-Dopa supplementation

Exclusion Criteria:

Patients should have been treated according to the Japanese insert slip

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Parkinson's disease patients in daily clinical settings
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2004-02; Primary Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (119):
- Japan (119):
  - Boehringer Ingelheim Investigational Site 11, Akita
  - Boehringer Ingelheim Investigational Site 95, Anan
  - Boehringer Ingelheim Investigational Site 1, Asahikawa
  - Boehringer Ingelheim Investigational Site 2, Asahikawa
  - Boehringer Ingelheim Investigational Site 26, Chiba
  - Boehringer Ingelheim Investigational Site 27, Chiba
  - Boehringer Ingelheim Investigational Site 60, Fuji
  - Boehringer Ingelheim Investigational Site 49, Fujisawa
  - Boehringer Ingelheim Investigational Site 25, Fukaya
  - Boehringer Ingelheim Investigational Site 103, Fukuoka
  - Boehringer Ingelheim Investigational Site 104, Fukuoka
  - Boehringer Ingelheim Investigational Site 105, Fukuoka
  - Boehringer Ingelheim Investigational Site 106, Fukuoka
  - Boehringer Ingelheim Investigational Site 56, Gifu
  - Boehringer Ingelheim Investigational Site 80, Habikino
  - Boehringer Ingelheim Investigational Site 3, Hakodate
  - Boehringer Ingelheim Investigational Site 59, Hamamatsu
  - Boehringer Ingelheim Investigational Site 64, Handa
  - Boehringer Ingelheim Investigational Site 82, Himeji
  - Boehringer Ingelheim Investigational Site 76, Hirakata
  - Boehringer Ingelheim Investigational Site 86, Hiroshima
  - Boehringer Ingelheim Investigational Site 87, Hiroshima
  - Boehringer Ingelheim Investigational Site 8, Ichinoseki
  - Boehringer Ingelheim Investigational Site 118, Kagoshima
  - Boehringer Ingelheim Investigational Site 15, Kamisu
  - Boehringer Ingelheim Investigational Site 50, Kashiwazaki
  - Boehringer Ingelheim Investigational Site 107, Kasuga
  - Boehringer Ingelheim Investigational Site 24, Kawagoe
  - Boehringer Ingelheim Investigational Site 46, Kawasaki
  - Boehringer Ingelheim Investigational Site 111, Kawatana
  - Boehringer Ingelheim Investigational Site 112, Kawatana
  - Boehringer Ingelheim Investigational Site 99, Kitakyushu
  - Boehringer Ingelheim Investigational Site 117, Kiyotake
  - Boehringer Ingelheim Investigational Site 83, Kobe
  - Boehringer Ingelheim Investigational Site 67, Koga
  - Boehringer Ingelheim Investigational Site 21, Koshiagya
  - Boehringer Ingelheim Investigational Site 63, Kōnan
  - Boehringer Ingelheim Investigational Site 12, Kōriyama
  - Boehringer Ingelheim Investigational Site 13, Kōriyama
  - Boehringer Ingelheim Investigational Site 100, Kurume
  - Boehringer Ingelheim Investigational Site 68, Kyoto
  - Boehringer Ingelheim Investigational Site 69, Kyoto
  - Boehringer Ingelheim Investigational Site 70, Kyoto
  - Boehringer Ingelheim Investigational Site 71, Kyoto
  - Boehringer Ingelheim Investigational Site 19, Maebashi
  - Boehringer Ingelheim Investigational Site 20, Maebashi
  - Boehringer Ingelheim Investigational Site 55, Matsumoto
  - Boehringer Ingelheim Investigational Site 88, Mihara
  - Boehringer Ingelheim Investigational Site 54, Minobu
  - Boehringer Ingelheim Investigational Site 116, Miyakonojō
  - Boehringer Ingelheim Investigational Site 114, Miyazaki
  - Boehringer Ingelheim Investigational Site 115, Miyazaki
  - Boehringer Ingelheim Investigational Site 77, Moriguchi
  - Boehringer Ingelheim Investigational Site 9, Morioka
  - Boehringer Ingelheim Investigational Site 23, Morohongō
  - Boehringer Ingelheim Investigational Site 53, Mukai-awagasaki
  - Boehringer Ingelheim Investigational Site 4, Muroran
  - Boehringer Ingelheim Investigational Site 51, Nagaoka
  - Boehringer Ingelheim Investigational Site 61, Nagoya
  - Boehringer Ingelheim Investigational Site 62, Nagoya
  - Boehringer Ingelheim Investigational Site 97, Nangōku
  - Boehringer Ingelheim Investigational Site 102, Naoetsu
  - Boehringer Ingelheim Investigational Site 28, Narita
  - Boehringer Ingelheim Investigational Site 93, Narutō
  - Boehringer Ingelheim Investigational Site 17, Nikkō
  - Boehringer Ingelheim Investigational Site 119, Nishihara
  - Boehringer Ingelheim Investigational Site 81, Nishinomiya
  - Boehringer Ingelheim Investigational Site 72, Osaka
  - Boehringer Ingelheim Investigational Site 98, Ōkawa
  - Boehringer Ingelheim Investigational Site 66, Ōtsu
  - Boehringer Ingelheim Investigational Site 108, Saga
  - Boehringer Ingelheim Investigational Site 45, Sagamihara
  - Boehringer Ingelheim Investigational Site 22, Saitama
  - Boehringer Ingelheim Investigational Site 79, Sakai
  - Boehringer Ingelheim Investigational Site 52, Sanjō
  - Boehringer Ingelheim Investigational Site 90, Sanyōonoda
  - Boehringer Ingelheim Investigational Site 5, Sapporo
  - Boehringer Ingelheim Investigational Site 6, Sapporo
  - Boehringer Ingelheim Investigational Site 7, Sapporo
  - Boehringer Ingelheim Investigational Site 110, Sasebo
  - Boehringer Ingelheim Investigational Site 78, Sayama
  - Boehringer Ingelheim Investigational Site 10, Sendai
  - Boehringer Ingelheim Investigational Site 91, Shimonoseki
  - Boehringer Ingelheim Investigational Site 18, Shimotsuke
  - Boehringer Ingelheim Investigational Site 85, Shingū
  - Boehringer Ingelheim Investigational Site 57, Shizuoka
  - Boehringer Ingelheim Investigational Site 58, Shizuoka
  - Boehringer Ingelheim Investigational Site 73, Suita
  - Boehringer Ingelheim Investigational Site 101, Tagawa
  - Boehringer Ingelheim Investigational Site 96, Takamatsu
  - Boehringer Ingelheim Investigational Site 74, Takatsuki
  - Boehringer Ingelheim Investigational Site 75, Takatsuki
  - Boehringer Ingelheim Investigational Site 109, Togitsu
  - Boehringer Ingelheim Investigational Site 92, Tokushima
  - Boehringer Ingelheim Investigational Site 30, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site 31, Tokyo Arakawa-ku
  - Boehringer Ingelheim Investigational Site 40, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 41, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 42, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 38, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site 32, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site 33, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site 43, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 39, Tokyo Nakano-ku
  - Boehringer Ingelheim Investigational Site 34, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 35, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 36, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site 37, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site 44, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site 113, Tomiai
  - Boehringer Ingelheim Investigational Site 14, Toride
  - Boehringer Ingelheim Investigational Site 65, Tsu
  - Boehringer Ingelheim Investigational Site 16, Tsukuba
  - Boehringer Ingelheim Investigational Site 29, Urayasu
  - Boehringer Ingelheim Investigational Site 84, Wakayama
  - Boehringer Ingelheim Investigational Site 89, Yamaguchi
  - Boehringer Ingelheim Investigational Site 47, Yokohama
  - Boehringer Ingelheim Investigational Site 48, Yokohama
  - Boehringer Ingelheim Investigational Site 94, Yoshinogawa

RESULTS

PARTICIPANT FLOW:
Groups:
- Pramipexole: BI-Sifrol® Tablets dose: 0.125 mg, 0.5 mg mode of administration: oral
Period: Overall Study
Arm/Group | Pramipexole
Started | 416
Completed | 188
Not Completed | 228
Not completed — Adverse Event | 49
Not completed — Lost to Follow-up | 88
Not completed — Withdrawal by Subject | 5
Not completed — Death | 6
Not completed — Lack of Efficacy | 13
Not completed — Physician Decision | 2
Not completed — No data was collected | 53
Not completed — Irregularly enrolled patients | 12

BASELINE CHARACTERISTICS:
Population: Data Set for Safety Analysis
Groups:
- Pramipexole: The number of patients enrolled was 416. The number of case report form which were collected was 364. Moreover the number of patients analyzed as safety analysis was 346 because 18 patients were excluded due to protocol violations.
Arm/Group | Pramipexole
Number analyzed (Participants) | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187
  Male | 159

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Adverse Events, Adverse Drug Reactions, Serious Adverse Events
Description: The aim of this Post Marketing Surveillance (PMS) was to obtain safety data in Parkinson's disease (PD) patients without concomitant use of levodopa for 3 years.
Time Frame: during 36 months
Population: 364 patients had available case report forms. Patients excluded: 5 patients with no visit since the first prescription, 12 irregularly enrolled patients, 9 excluded from analysis according to regulatory requirement, and 1 patient with no safety data available. As a result, there were 346 patients in the safety analysis set.
Measure: Number; unit: Proportion (percentage of participants)
Groups:
- Pramipexole: Substance (INN): Pramipexole Trade name: BI-Sifrol® Pharmaceutical form: Tablet Source: Marketed products (There was no investigational products in this PMS) Unit strength: 0.125 mg and 0.5 mg Daily dose: Approved dose range (From 0.25 mg/day to 4.5 mg/day) Duration of use: 3 years Route of administration: Orally
Arm/Group | Pramipexole
Number analyzed (Participants) | 346
Proportion (percentage of participants)
  Proportion of Adverse Events | 51.7
  Proportion of Adverse Drug Reactions | 41.3
  Proportion of Serious Adverse Events | 8.4

2. Secondary Outcome: Clinical Global Impression of Improvement
Description: Investigators evaluation of the PD symptoms on a rating scale of 5 categories (very much improved, much improved, minimally improved, no effect, and unassessable).
Time Frame: after 36 months treatment
Population: There were 346 patients in the safety analysis set. Patients excluded from this population: 5 because of administration to patients who didn't suffer from PD and 2 with no efficacy data available. As a result, 339 patients were evaluated for efficacy.
Measure: Number; unit: Participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 339
Participants
  Very much improved | 19
  Much improved | 137
  Minimally improved | 97
  No effect | 15
  Unassessable | 71

3. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score
Description: Motor examination is assessed by 27 questionnaire items in UPDRS Part III section. Each item is scored from 0 (best) to 4 (worst), and the total score of UPDRS Part III is from 0 (best) to 108 (worst). A decrease in the score means improvement.
Time Frame: Baseline and at 36 months (or at the time of discontinuation)
Population: The number of patients (291) means a population who have the assessment of UPDRS Part III total score at baseline and at least one post-visit after administration of pramipexole.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 291
Unit on a scale | -5.2 (11.2)

4. Secondary Outcome: Change From Baseline in Modified Hoehn & Yahr Rating Scale
Description: A severity of PD symptom are assessed by Modified Hoehn & Yahr rating scale. This scale consist of 10 levels including additional evaluation levels defined in Japan. Ten levels are described by 0 (best), 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5 (worst).
Time Frame: Baseline and at 36 months (or at the time of discontinuation)
Population: The number of patients (295) means a population who have the assessment of Modified Hoehn & Yahr rating scale at baseline and at least one post-visit after administration of pramipexole.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 295
Unit on a scale | -0.1 (0.7)

ADVERSE EVENTS:
Time Frame: 36 months
Groups:
- Pramipexole: The drug was administered orally to patients according to the package insert in Japan. The drug form is only tablet. The initial dose was 0.125 mg twice a day, and was escalated in case of lack of efficacy. The maintenance dose was between 1.5 mg/day and 4.5 mg/day (0.5 mg - 1.5 mg three times a day).
Arm/Group | Pramipexole
Serious Adverse Events (participants affected / at risk) | 29/346
Other Adverse Events (participants affected / at risk) | 106/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=346)
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Agitation (Psychiatric disorders) | 1
Delusion (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Diabetic hyperosmolar coma (Nervous system disorders) | 1
Neuroleptic malignant syndrome (Nervous system disorders) | 2
Thalamus haemorrhage (Nervous system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Death (General disorders) | 1
Hernia (General disorders) | 1
Pyrexia (General disorders) | 1
C-reactive protein increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=346)
Hallucination (Psychiatric disorders) | 28
Somnolence (Nervous system disorders) | 59
Constipation (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.